CLINICAL TRIAL: NCT02815631
Title: Assessing the Efficacy of CARDIOgoniometry (CGM) to Determine Physiologically Significant Stenosis in Patients With Stable Coronary Artery Disease in Comparison to Fractional FLOW Reserve - CARDIOFLOW
Acronym: CARDIOFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 15/YH/2071
Record Dates: First submitted 2016-02-18; First posted 2016-06-28 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease
Keywords: fractional flow reserve; cardiogoniometry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiogoniometry (CGM) (Experimental): Every patient involved in the study will undergo a series of CGM recordings whilst having their FFR procedure. These recordings will all be done whilst they are in the catheterisation laboratory and will be taking at the following points during the procedure.
  1. First baseline recording - taken when the patient first enters the catheterisation laboratory and is prepped for their procedure.
  2. Second baseline recording - taken when the FFR guide wire is in place in the coronary artery being assessed.
  3. Maximal hyperaemia recording - this will be taken when the patient is at maximal hyperaemia during their adenosine infusion for their FFR procedure.
  The patients involvement will then be finished in the study and will be cared for as per clinical practice.
  If the CGM records a result of anything less than 0, it will be regarded as a positive result.
  Interventions: Device: Cardiogoniometry (CGM)
- Fractional flow reserve (FFR) (Active Comparator): Every patient involved in the study will undergo an FFR assessment of their coronary arteries. These recordings will all be done whilst they are in the catheterisation laboratory. They will have the following recordings:
  1. A baseline FFR will be recorded once the pressure wire has been advanced down the coronary artery being assessed.
  2. Maximal hyperaemia FFR will be recorded during adenosine infusion.
  An FFR ratio of <0.80 will be regarded as a positive result.
  Interventions: Device: Fractional Flow Reserve (FFR)

INTERVENTIONS:
Device: Cardiogoniometry (CGM)
  Arms: Cardiogoniometry (CGM)
Device: Fractional Flow Reserve (FFR)
  Arms: Fractional flow reserve (FFR)

SUMMARY:
The CARDIOFLOW study compares the standard test, a pressure wire test called fractional flow reserve (FFR), with a new method that is based on taking a detailed "3D" ECG called Cardiogoniometry (CGM).

FFR is an angiographic technique which measures the physiological significance of a coronary stenosis and trial data has shown that basing management decisions on this data improves prognosis. However FFR studies are expensive and invasive, whereas CGM is painless and simply involves placing 4 sticky pads to the patient's chest / back and is similar to an ECG (heart tracing). The investigators want to see whether we can use this new method to find out whether treatment with coronary angioplasty would be of benefit. If so, then in the future, clinicians could use this method (CGM) rather than pressure wire assessment (FFR). This would have several advantages; in particular, it can be easily performed in the clinic and avoids the need to use an expensive pressure wire.

DETAILED DESCRIPTION:
This study aims to test the hypothesis that cardiogoniometry (CGM) is helpful to identify physiologically significant coronary artery stenosis in comparison to fractional flow reserve (FFR).

Last year in the UK 202 098 patients underwent coronary angiography to determine whether they had significant coronary artery disease. However, it is well recognised that, even with orthogonal views, angiography is limited in terms of its ability to determine the functional importance of coronary lesions. In particular those lesions judged to be 50-70% stenosed may not necessarily cause ischaemia as this depends on factors such as the lesion length and, importantly, the size of the territory supplied by the vessel.

There have been several studies that have demonstrated the clinical utility of evaluating such lesions with FFR. The measurement of FFR is an index of the physiological significance of a coronary stenosis and is defined as the ratio of maximal blood flow in a stenotic artery to normal maximal flow. It is calculated by comparing the ratio of the aortic pressure and the pressure distal to the coronary stenosis during maximal hyperaemia. These pressures are measured by introducing a coronary pressure guide wire into the artery and hyperaemia is induced by giving an infusion of adenosine intravenously. An FFR ratio of <0.80 indicates that the coronary stenosis is causing significant ischaemia and would benefit from PCI. This has since been incorporated into ESC clinical guidelines on myocardial revascularisation.

However this is an invasive procedure and the pressure wires are relatively expensive compared to standard angioplasty wires. On the contrary, CGM is a cheap and non-invasive technique that can be easily applied. The aim of the proposed study is to assess whether CGM may be able to aid clinicians in identifying if a coronary stenosis is physiologically significant at inducing myocardial ischaemia in conjunction with standard coronary angiography.

CGM is form of 3D vector electrocardiography which can provide quantitative analysis of myocardial depolarisation and repolarisation. It has been shown to be more sensitive and specific than standard 12-lead ECG at diagnosing stable coronary artery disease. Furthermore, other work has showed CGM to be more sensitive than 12-lead ECG at detecting patients with ACS. More recently in 2012, further work found that CGM was more sensitive and specific than the 12 lead ECG at identifying abnormal myocardial perfusion scans (MPS). FFR validity was initially based on a comparison with MPS and therefore we hypothesise that CGM may be comparable to FFR.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with stable coronary artery disease for elective percutaneous coronary intervention (PCI)
* Patients who have been consented to undergo coronary angiography +/- PCI as part of their routine care by their clinician.
* Aged 18 or over.
* The patient has been informed of the nature of the study and has provided full written informed consent.
* FFR will be performed on study participants who demonstrate visible coronary stenosis on coronary angiography.

Exclusion Criteria:

* Patients unable to give informed consent including those with communication difficulties due to poor English.
* Patients with haemodynamic instability and / or cardiogenic shock (defined as a sustained blood pressure of <90mmHg +/- the need for inotropic support)
* Patients with an acute coronary syndrome (as defined by the European Society of Cardiology)
* Those unable to perform a good quality CGM: 1) Patients who are SOB at rest; 2) Patients with very frequent ectopic beats; 3) Patients in atrial fibrillation; 4) Patients with a heart rate >150 beats/min
* Those patients unable to tolerate adenosine: 1) Patients with severe asthma, especially if taking oral theophylline; 2) Patients with second or third degree heart block (without a pacemaker in situ); 3) Patients with sick sinus syndrome; 4) Patients with Long QT syndrome; 5)Patients with severe hypotension (systolic pressure) <100mmHg); 6) Patients with decompensated heart failure.
* Patients with previous coronary artery bypass graft surgery
* Patients who are unable to receive treatment with heparin
* Patients with a chronic total occlusion
* Patients with extremely tortuous or calcified vessels that are unfavourable for assessment with FFR.
* Patients with severe stenosis of the left main stem
* Patients with significant renal impairment (defined as eGFR<30ml/min)
* Females who are or could be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of CGM to detect physiologically important coronary stenosis. | Calculated within 30 days after participant recruitment is complete.
  The sensitivity of CGM to detect physiologically important coronary stenosis will be calculated after all participants are recruited. The number of patients which had true positive results (that is CGM tested positive when they had significant coronary disease) will be divided by the total number of participants who were found to have physiologically important coronary stenosis and expressed as a percentage
Specificity of CGM to detect physiologically important coronary stenosis | Calculated within 30 days after participant recruitment is complete.
  The specificity of CGM to detect physiologically important coronary stenosis will be calculated after all participants are recruited. The number of patients which had true negative results (that is CGM tested negative when they did not have significant coronary disease) will be divided by the total number of participants who were found not to have physiologically important coronary stenosis and expressed as a percentage.
Positive predictive value (PPV) of CGM to detect physiologically important coronary stenosis | Calculated within 30 days after participant recruitment is complete.
  The PPV of CGM to detect physiologically important coronary stenosis will be calculated after all participants are recruited. The number of patients which had true positive results (that is CGM tested positive when they had significant coronary disease) will be divided by the total number of participants who had a positive CGM test and expressed as a percentage.
Negative predictive value (NPV) of CGM to detect physiologically important coronary stenosis | Calculated within 30 days after participant recruitment is complete.
  The NPV of CGM to detect physiologically important coronary stenosis will be calculated after all participants are recruited. The number of patients which had true negative CGM result (that is CGM tested negative when they didn't not have significant coronary disease) will be divided by the total number of participants who had a negative CGM result and expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Hull, East Yorkshire, United Kingdom

REFERENCES:
- [Result] Brown OI, Clark AL, Chelliah R, Davison BJ, Mather AN, Cunnington MS, John J, Alahmar A, Oliver R, Aznaouridis K, Hoye A. Cardiogoniometry Compared to Fractional Flow Reserve at Identifying Physiologically Significant Coronary Stenosis: The CARDIOFLOW Study. Cardiovasc Eng Technol. 2018 Sep;9(3):439-446. doi: 10.1007/s13239-018-0354-1. Epub 2018 Apr 12. PMID 29651685
- See also: Cardiogoniometry Compared to Fractional Flow Reserve at Identifying — https://link.springer.com/article/10.1007%2Fs13239-018-0354-1